CLINICAL TRIAL: NCT01161303
Title: Study to Investigate the Role of TNF-alpha in Asthma Using Biopsy Explants and Primary Bronchial Epithelial Cell Cultures
Brief Title: An Investigation of Tumor Necrosis Factor (TNF)-Alpha in Asthma Using Biopsy Explants and Primary Bronchial Epithelial Cell Cultures
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Professor S.T. Holgate, University of Southampton
Other Study IDs: SUHT-III-KSB
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Asthma
Keywords: Asthma; TNF alpha; epithelial cell culture
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * bronchial brushings and biopsies
  * Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
We have developed in vitro systems including primary epithelial cell cultures and explant cultures of bronchial tissues to study the interaction between the bronchial mucosa and allergens. This approach involves culturing bronchial biopsies under optimal conditions and stimulate them with allergens thus enabling us to perform a dynamic study without the need of performing several bronchoscopies and will allow the testing of unapproved substances, which could, otherwise, not be delivered, in vivo.

We wish to apply these ex vivo bronchial culture systems to assess cytokine release in moderately severe asthmatics and evaluate the effects of blocking TNF-alpha signalling using anti TNF-alpha monoclonal antibodies.

DETAILED DESCRIPTION:
Volunteers with moderately severe asthma will be recruited and carefully characterized in terms of lung function, asthma symptom scores, medication usage and allergen sensitivity (by blood and skin tests). If suitable, they will then be asked to withdraw their corticosteroids for a week with careful monitoring of the symptoms and peak flows before undergoing fibreoptic bronchoscopy as was carried out in the previous explant study. Bronchial brushings and biopsies will be carried out as per standard technique used in University medicine. Primary epithelial cell cultures will be established from bronchial brushings and will be used for optimising the dose of anti TNF-alpha required for inhibition of TNF-alpha induced responses. The biopsies will be placed in either culture medium alone, allergen extract or allergen extract plus anti TNF-alpha antibody and cultured for 24 hours. The biopsies will then be either snap frozen in liquid nitrogen for analysis of cytokines or processed for immunohistochemical analysis. The supernatants from each study will be recovered and analysed for cytokine (IL-5, IL-8, IL-13, MIP 1 alpha and RANTES) release by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Moderately severe asthmatics
* Male or female
* Uses inhaled beclomethasone 400-1000 mcg or equivalent
* Documented positive skin test to common allergens and
* FEV1 of >60% predicted

Exclusion criteria:

* Smokers
* Subjects with an acute asthmatic episode in the last 6 weeks
* Other significant clinical illnesses
* Pregnant women
* Those sensitive to lignocaine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2000-07; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T Holgate, MD, Principal Investigator — University of Southampton
Locations (1):
- Southampton University Hospital Trust, Southampton, Hampshire, United Kingdom

REFERENCES:
- [Result] Babu KS, Puddicombe S, Shaw TJ, Howell T, Wilson SJ, Holgate ST, Davies DE. Am J Respir Crit Care Med. 169 (7): A801, 2004